CLINICAL TRIAL: NCT01801800
Title: Speckle Tracking Assessment of Cardiac Function in Severe Aneurysmal Subarachnoid Haemorrhage and Impact on Neurologic Outcome (SPLASH)
Brief Title: Cardiac Function in Severe Aneurysmal Subarachnoid Haemorrhage Patients
Acronym: SPLASH
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0410
Record Dates: First submitted 2013-02-15; First posted 2013-03-01 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Aneurysmal Subarachnoid Haemorrhage; World Neurosurgeon Federation Score ≥ III
Keywords: Aneurysmal subarachnoid haemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aneurysmal subarachnoid haemorrhage: Speckle-tracking images in Echocardiography
  Interventions: Procedure: Echocardiography

INTERVENTIONS:
Procedure: Echocardiography — Speckle-Tracking of echocardiographic loops by a cardiologist blinded to the patient's management and outcome

SUMMARY:
Cardiac dysfunction can occur in aneurysmal subarachnoid haemorrhage and might impact patient's neurologic outcome Condition Aneurysmal subarachnoid haemorrhage World Neurosurgeon Federation Score ≥ III

DETAILED DESCRIPTION:
Trans-thoracic echocardiography on day 1, day 3 and day 7 Speckle-Tracking of echocardiographic loops by a cardiologist blinded to the patient's management and outcome

ELIGIBILITY:
Inclusion Criteria:

* Aneurysmal subarachnoid haemorrhage
* World Neurosurgeon Federation Score ≥ III
* Written information to next-of-kin and patients when possible

Exclusion Criteria:

* History of myocardial infarction, chronic heart failure with NYHA ≥ 2, major heart surgery
* Lack of acoustic window to perform trans-thoracic echocardiography

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe Aneurysmal subarachnoid haemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Neurologic outcome | 3 months
  modified Rankin Scale (mRS). Poor neurological outcome was considered as death or severe disability (mRS 5-6).

SECONDARY OUTCOMES:
Correlation between cardiac strain on day 1 and Left Ventricular Ejection fraction | Day 1
Correlation between cardiac enzymes (NT-proBNP, troponin T US) and cardiac strain | Day 1
Correlation between EKG findings and cardiac strain | Day 1
Time to amines discontinuation | During Intensive Care Unit stay, expected average 17 days
Duration of mechanical ventilation | Duration of mechanical ventilation, expected average 15 days
Length of ICU stay | Duration of ICU stay, expected average 17 days
Correlation between Cardiac function and Mechanical Ventilation | Day1, day3, day7 and extubation time expected average 15 days
Correlation between Cardiac function and ICU length of stay | Day1, day3, day 7 and end of stay in ICU expected average 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Cinotti, MD, Principal Investigator — Nantes University Hospital; Bertrand ROZEC, PhD, MD, Study Chair — Nantes University Hospital
Locations (2):
- France (2):
  - University Hospital, Nantes
  - University Hospital, Rennes

REFERENCES:
- [Background] Hofmeijer J, Kappelle LJ, Algra A, Amelink GJ, van Gijn J, van der Worp HB; HAMLET investigators. Surgical decompression for space-occupying cerebral infarction (the Hemicraniectomy After Middle Cerebral Artery infarction with Life-threatening Edema Trial [HAMLET]): a multicentre, open, randomised trial. Lancet Neurol. 2009 Apr;8(4):326-33. doi: 10.1016/S1474-4422(09)70047-X. Epub 2009 Mar 5. PMID 19269254